CLINICAL TRIAL: NCT05969301
Title: Role of the Memory in the Spinal Exercises for Adolescent Idiopathic Scoliosis
Brief Title: Memory and Scoliosis Spinal Exercises
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: International Institute of Behavioral Medicines (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-003
Record Dates: First submitted 2023-07-16; First posted 2023-08-01 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Health-related quality of life; Adolescents; Memory; Scoliosis; Exercise
MeSH Terms: conditions — Scoliosis; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Specific spinal exercises for idiopathic scoliosis — The spinal esercises mainly include: active self-correction, strengthening spinal deep muscles while maintaining self-correction, segmentary stretching involving the limbs and back muscles, and postural task-oriented exercises (e.g. walking, standing, sitting).

SUMMARY:
This is a behavioral observational study aimed at evaluating the impact that spinal exercises exert on memory of young people. It consists of a short self-administered questionnaire which will be given to adolescents with scoliosis to complete. Relationships between young individuals' answers and health-related quality of life will be evaluated.

DETAILED DESCRIPTION:
This is a behavioral observational study aimed at evaluating the impact that spinal exercises exert on memory of young people. Literature found out that a memory-experience difference exists between pleasant and unpleasant situations and young people are expected to capture memories more accurately when these, as voiced for instance by outcome measures of health-related quality of life, are at their worst- rather than at their best-perceived level.

In Literature there are not studies which investigate the relationships between the memory of spinal exercises as for adolescents with idiopathic scoliosis and health-related quality of life.

The study consists of a short self-administered questionnaire which will be given to young persons to complete. In more details, the survey is made of four questions collecting information on time to learn an exercise, time to perform an exercise, difficulty to do the exercise, commitment to perform the exercise. Further, participants will have to complete a self-administered health-related quality of life questionnaire, and namely the Scoliosis Research Society-22 patients questionnaire.

Descriptive statistics will be presented by taking into account the socio-demographic characteristics of the sample being investigated. Statistical correlations between adolescents' answers and health-related quality of life questionnaire will be also evaluated.

This study's usefulness relies on understanding which spinal exercises impact more on memory in order to increase a young persons' positive routines and improve their performance with rehabilitative programs, with the ultimate goal of growing their adherence to and satisfaction with treatment.

ELIGIBILITY:
Inclusion Criteria:

* a primary diagnosis of Adolescent Idiopathic Scoliosis determined by expert clinicians
* ability to read and understand the Italian language

Exclusion Criteria:

* any diagnosable cause of scoliosis
* leg-length discrepancy of > 1 cm
* lower limb deformities interfering with spinal posture,
* cardiac and/or respiratory dysfunction
* systemic illness
* previous spinal surgery,
* cognitive impairment
* refusal to adhere to the study

Ages: 11 Years to 19 Years | Sex: All
Age Groups: Child, Adult
Study Population: Adolescent idiopathic scoliosis, which is a three-dimensional deformity of the spine and trunk occurring in healthy pubertal children.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-02-29 (Estimated); Study Completion 2024-02-29 (Estimated)

PRIMARY OUTCOMES:
SRS-22 patient questionnaire | At the moment of the assessment
  Scoliosis Research Society-22 patient questionnaire. The maximum score in each domain (pain, function, self-image, and mental health) is 5 and minimum score is 1, with higher scores representing greater individual's quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Barbara Rocca, Calosso, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Monticone M, Ambrosini E, Cazzaniga D, Rocca B, Ferrante S. Active self-correction and task-oriented exercises reduce spinal deformity and improve quality of life in subjects with mild adolescent idiopathic scoliosis. Results of a randomised controlled trial. Eur Spine J. 2014 Jun;23(6):1204-14. doi: 10.1007/s00586-014-3241-y. Epub 2014 Feb 28. PMID 24682356
- [Result] Monticone M, Baiardi P, Calabro D, Calabro F, Foti C. Development of the Italian version of the revised Scoliosis Research Society-22 Patient Questionnaire, SRS-22r-I: cross-cultural adaptation, factor analysis, reliability, and validity. Spine (Phila Pa 1976). 2010 Nov 15;35(24):E1412-7. doi: 10.1097/BRS.0b013e3181e88981. PMID 21030889